CLINICAL TRIAL: NCT05253482
Title: Efficacy of Wet Cupping Therapy on Fibromyalgia Syndrome a Randomised Controlled Trial
Brief Title: Efficacy of Wet Cupping Therapy on Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Training consultant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCT 7
Record Dates: First submitted 2022-02-09; First posted 2022-02-23 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Fibromyalgia
Keywords: wet cupping therapy; fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will undergo 3 successive wet cupping therapy (WCT) sessions once in a month throughout 3 months (On 0, 30, and 60 days
  Interventions: Procedure: wet cupping therapy
- Control group (No Intervention): Control group will not receive any intervention

INTERVENTIONS:
Procedure: wet cupping therapy — Vacuum cups will used on different acupuncture points to perform WCT: The one on the posterior median line, in the depression below the processus spinosus of the 7th cervical vertebra was DU 14 (Dazhui) point; the ones on the back, 3.0 cm lateral to the lower border of the spinous process of the 3rd thoracic vertebra interscapulum region were UB 42 (Pohu) bilateral points; and the ones on the back, 3.0 cm lateral to the lower border of the spinous process of the 7th thoracic vertebra were UB 46 (Geguan) bilateral points and additionally the patient's trigger points which we detect during the examination. There will be 5-7 points in total. The technique used will be triple S (Sucking, Scarification, Sucking) in all sessions.
  Arms: Intervention group

SUMMARY:
Background and purpose: Although wet cupping therapy (WCT) is in use, clinical investigations of its efficiency are scarce. The aim of this study was to evaluate the effects of wet cupping therapy (WCT) on fibromyalgia syndrome Methods: The patients will be randomized into two groups. WCT will be applied once a month to patients in the intervention group while the control group will be on standard therapy for fibromyalgia. An evaluation will be made before treatment and at the 3rd month using the Fibromyalgia Impact Survey (FEA), VAS, and EuroQol-5D (EQ-5D-3L) quality of life scale.

DETAILED DESCRIPTION:
Background: Cupping therapy is a traditional treatment method especially belonging to our geography. In addition to being on the agenda as a traditional treatment method all over the world in recent years, it has also been the subject of an increasing number of scientific studies in the medical literature. In addition to studies investigating positive effects on blood biochemistry such as reducing LDL and TGS levels (1,2), removing heavy metals from the blood (3), there are also studies showing that it is effective in the treatment of migraine (4) and in the treatment of nonspecific low back pain (5). As a result of clinical studies, it was determined that cupping is effective in painful conditions (headache, myofascial pain, fibromyalgia), calcification, gonorrhea, spondylosis.

It has also been found to be effective in skin diseases (such as acne, herpes zoster), vascular diseases, blood pressure problems, lung and respiratory diseases, and some psychiatric disorders (as a tranquilizer in depression, schizophrenia)(6,7,8,9,10,11, 12,13). It has been suggested that wet cupping therapy stimulates healing by removing inflammatory mediators and toxins from the body. Some practitioners claim that it reduces or even seizes pain by regulating the autonomic nervous system. (13).

Purpose: The aim of our study is to investigate how and to what extent wet cupping therapy will affect the patients diagnosed with fibromyalgia.

Method: The patients who were referred to Umraniye Training Hospital Physical Therapy and Rehabilitation Polyclinic will be enrolled in the study.

The inclusion criteria are being 18-65 years old, having been diagnosed with fibromyalgia (ACR 2016 diagnosis criteria), and consenting to participate in the study. Those who are accompanied with any chronic disease and on daily medication, contraindicated to WCT as determined in the routine blood tests that were routinely performed before the prior to application (Hgb <9,5; INR> 1,2,; Hgb <9,5, etc) and who received WCT in the last three months will be excluded.

The volunteers will be randomized into two separate groups as study and control group Control group will not receive any intervention while the study group will undergo 3 successive WCT sessions once in a month throughout 3 months (On 0, 30, and 60 days). Vacuum cups will used on different acupuncture points to perform WCT: The one on the posterior median line, in the depression below the processus spinosus of the 7th cervical vertebra, was DU 14 (Dazhui) point; the ones on the back, 3.0 cm lateral to the lower border of the spinous process of the 3rd thoracic vertebra interscapulum region were UB 42 (Pohu) bilateral points; and the ones on the back, 3.0 cm lateral to the lower border of the spinous process of the 7th thoracic vertebra were UB 46 (Geguan) bilateral points and additionally the patient's trigger points which we detect during the examination. There will be 5-7 points in total. The technique used will be triple S (Sucking, Scarification, Sucking) in all sessions.

At 0 and 3 months, to both patient groups those questionnaires: Fibromyalgia Impact Survey (FEA), VAS, and EuroQol-5D (EQ-5D-3L) quality of life scale will be applied. Evaluation will be made between two groups regarding the scores of those scales

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are being 18-65 years old, having been diagnosed as fibromyalgia (ACR 2016 diagnosis criteria) and consenting to participate in the study

Exclusion Criteria:

* Those who are accompanied with any chronic disease and on daily medication, contraindicated to WCT as determined in the routine blood tests that were routinely performed before the prior to application (Hgb <9,5; INR> 1,2,; Hgb <9,5, etc) and who received WCT in the last three months will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline (at 0 month) Fibromyalgia Impact Questionnaire (FIQ) scores at 3 month | At 0 and 3 months
  This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week.

SECONDARY OUTCOMES:
Change from baseline EuroQol-5D (EQ-5D-3L) quality of life scale scores at 3 month. | At 0 and 3 months
  The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change from baseline (At 0 month) Visual Analog Scale (VAS) scores at 3 month | At 0 and 3 months
  VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Emin Pala, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)